CLINICAL TRIAL: NCT01080326
Title: Feasibility of Translumenal Endoscopic Omental Patch Closure of Perforated Viscus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Natural Orifice Surgery Consortium for Assessment and Research (Other)
Responsible Party: Principal Investigator, Juliane Bingener-Casey, PI, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 08-008389; ULIRR024150 (Other Grant/Funding Number: NOSCAR)
Record Dates: First submitted 2010-03-02; First posted 2010-03-04 (Estimated); Results first posted 2015-04-14 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Peptic Ulcer
Keywords: ulcer repair surgery; transluminal omental patch
MeSH Terms: conditions — Peptic Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Endoscopic Translumenal Omental Patch (Experimental): Patients with the clinical diagnosis of a perforated viscus who are scheduled to undergo surgical exploration will be recruited. The endoscope will be gently advanced through the ulcer. Irrigation with saline will proceed. Then a viable mobile piece of omentum will be identified and pulled into the ulcer. After the omentum is located in the stomach, clips will be used to fix the Endoscopic Translumenal Omental Patch in place.
  Interventions: Device: Endoscopic Translumenal Omental Patch

INTERVENTIONS:
Device: Endoscopic Translumenal Omental Patch — The endoscope will be gently advanced through the ulcer. Irrigation with saline will proceed. Then a viable mobile piece of omentum will be identified and pulled into the ulcer. After the omentum is located in the stomach, clips will be used to fix it in place.
  Other Names: Ulcer repair surgery

SUMMARY:
This study is being done to see if a new approach to repair perforated ulcers in the stomach (holes in the stomach) or the first part of the intestine is possible. Traditionally, either open operations (large single incision) or laparoscopic operations (multiple small camera-guided incisions) have been used to repair perforated ulcers. Over the last ten years, some surgeons have used endoscopic equipment to assist them with performing the procedure. It is unknown if perforated ulcer repair can be done using an endoscope as the main instrument (a flexible tube with a video camera inserted into the stomach through your esophagus) to "patch" or plug the perforation. We will patch the perforation using a standard method which uses tissue from outside the stomach. A laparoscopic camera will also be used to assist our view. This study is intended to be a feasibility study to demonstrate the endoscopic technique can be safely performed

Hypothesis: The primary outcome is successful completion of the procedure.

DETAILED DESCRIPTION:
Perforation is the most dangerous complication of gastroduodenal ulcer disease. It accounts for more than 70% of deaths associated with peptic ulcer disease. In addition to age and concomitant disease, intervention related complications are statistically significant predictors of death after hospital stay. Age, time to presentation and comorbidities are not factors that can be influenced. If it would be possible to reduce the impact of procedure related complications or the "second hit", that may lead to decreased morbidity and mortality.

This will be a pilot clinical study to evaluate the safety and feasibility of endoscopic translumenal omental patch closure. Patients with the clinical diagnosis of a perforated viscus who are scheduled to undergo surgical exploration will be recruited. Endoscopic translumenal omental patch will be attempted first if the patient has no contraindication. Should this prove unsuccessful, the surgical team will proceed with conversion to laparoscopic or open standard surgical therapy as indicated.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with clinical diagnosis of a perforated viscus who are scheduled to undergo surgical intervention
* Surgical candidate for endoscopic, laparoscopic, or open procedure
* Age > 21
* Informed written consent

Exclusion Criteria:

* Prior gastric or duodenal surgery
* Prior total abdominal colectomy or transverse colectomy
* Prior omentectomy or omental flaps
* Known perforation site other than stomach or duodenum
* Patients with contra-indications for laparoscopy
* Patients with contraindications for endoscopy
* Upper gastrointestinal anatomy that would preclude endoscopic therapy
* Coagulopathy or thrombocytopenia
* Pregnant patients
* Patients <21 years of age
* Prisoners
* Patients found at surgery to have disease processes other than perforated peptic ulcer disease will be asked for permission to record their data for comparison

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juliane Bingener-Casey, MD.S, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Bingener J, Loomis EA, Gostout CJ, Zielinski MD, Buttar NS, Song LM, Baron TH, Ghahfarokhi LS, Rajan E. Feasibility of NOTES omental plug repair of perforated peptic ulcers: results from a clinical pilot trial. Surg Endosc. 2013 Jun;27(6):2201-8. doi: 10.1007/s00464-012-2740-3. Epub 2013 Jan 26. PMID 23355151

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled between February 2010 and February 2012 at Mayo Clinic in Rochester, Minnesota.
Period: Overall Study
Arm/Group | Endoscopic Translumenal Omental Patch
Started | 7
Completed | 3
Not Completed | 4
Not completed — Patient deterioration prior to procedure | 3
Not completed — Surgeon decision | 1

BASELINE CHARACTERISTICS:
Population: This includes only those participants for whom ulcer repair was attempted. Participants who were excluded in the operating room (OR) for previously unknown complications were not included.
Arm/Group | Endoscopic Translumenal Omental Patch
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Completing Natural Orifice Translumenal Endoscopic Surgical (NOTES) Repair
Description: At the time of surgery the repair was pressure tested using endoscopic insufflation. Two days post-operation all participants receiving the NOTES repair underwent a water-soluble contrast study to demonstrate leakage.
  Note: The NOTES procedure was attempted first if the subject had no contraindication. If this proved unsuccessful the surgical team proceeded with conversion to laparoscopic or open standard surgical therapy as indicated.
Time Frame: 2 days post-operation
Measure: Number; unit: participants
Arm/Group | Endoscopic Translumenal Omental Patch
Number analyzed (Participants) | 3
participants
  Participants completing NOTES repair | 2
  Participants completing other procedure | 1

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Endoscopic Translumenal Omental Patch
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endoscopic Translumenal Omental Patch (N=3)
Colotomy (Gastrointestinal disorders) | 1 (1) — Conversion to open procedure was necessary, as a laparoscopic repair was deemed not feasible. After laparotomy, a colotomy in the transverse colon was encountered.
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Subject has long history of chronic obstructive pulmonary disease (COPD), received upper midline incision for non-study portion of procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes